CLINICAL TRIAL: NCT00518115
Title: A 16-Week, Parallel-Group, Double-Blind, Randomized, Placebo-Controlled, Multicenter, Dose-Ranging Study to Evaluate the Efficacy, Safety, and Tolerability of Multiple Doses and Multiple Treatment Regimens of GSK716155, With Byetta as an Open Label Active Reference, in Subjects With Type 2 Diabetes Mellitus
Brief Title: Out-Patient Study in Patients With Type 2 Diabetes Mellitus Who Are Taking no Diabetes Medication or Metformin Only
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GLP110125
Record Dates: First submitted 2007-08-17; First posted 2007-08-20 (Estimated); Results first posted 2014-06-23 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: GLP-1,; Type 2 Diabetes,; pharmacokinetics,; pharmacodynamics,; GSK716155,; metformin,; exenatide; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — rGLP-1 protein; Exenatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Albiglutide (GSK716155) or exenatide — Albiglutide weekly subcutaneous injection or exenatide twice daily injection

SUMMARY:
This study is a placebo-controlled study in patients with Type 2 Diabetes Mellitus who are either taking no diabetes medication or who are taking metformin only. This study will investigate the safety, tolerability, and efficacy of Albiglutide (GSK716155) and will measure the levels of Albiglutide (GSK716155) in the bloodstream when it is given for 16 weeks. As a comparison, some subjects will receive exenatide instead of Albiglutide (GSK716155). The study will involve weekly visits for 17 weeks,and less frequent follow-up visits for an additional 10 weeks. Assessments include repeat blood sampling and monitoring of any side effects.

DETAILED DESCRIPTION:
A 16-week, parallel-group, double-blind, randomized, placebo-controlled, multicenter, dose-ranging study to evaluate the efficacy, safety and tolerability of multiple doses and multiple treatment regimens of Albiglutide (GSK716155) with Byetta as an open-label active reference, in subjects with Type 2 Diabetes Mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Has type 2 diabetes mellitus as defined by the criteria of the American Diabetes Association and recognized by World Health Organization Expert Committee on the Diagnosis and Classification of Diabetes Mellitus [American Diabetes Association, 2004a] at least three months preceding screening
* Has concurrent type 2 diabetes mellitus therapy: Must be diet and exercise treated; must not have taken antidiabetic medication for at least three months prior to prescreening or Monotherapy with metformin, with a history of a stable dose for at least three months before prescreening (not taking more than one oral antidiabetic agent)
* Has HbA1c level at screening ≥7 and ≤10%
* Is male or female 18 to 75 years of age, inclusive, at screening
* Has body mass index ≥20 and ≤40 kg/m²
* If subject is a smoker, must be able to abstain while in clinic at each visit
* If female, is eligible to enter and participate throughout the study, including the follow-up period: 1) If of nonchildbearing potential (i.e. physiologically incapable of becoming pregnant {tubal ligation}, including any female who is postmenopausal [>1 year without menstrual period]); or, 2) If of childbearing potential, has negative pregnancy tests at screening (serum) and at baseline (urine) and: 3) Has a male partner who is sterile prior to the female subject's entry into the study and is the sole sexual partner for that female subject, or 4) Uses double-barrier methods of contraception; condoms (with spermicide) and intrauterine devices are acceptable, or 5) Uses hormonal contraceptives (oral, depots, patches, etc) with double-barrier methods of contraception as outlined above, or, 6) Abstains from sexual intercourse, or 7) Is with a same-sex partner and does not participate in bisexual activities where there is any risk of pregnancy
* Signs and dates informed consent before any study-related procedures are performed

Exclusion Criteria:

* Has metabolic disease including but not limited to: 1) Diagnosis of type 1 diabetes mellitus, 2) Uncorrected thyroid dysfunction (NOTE: subjects with hypothyroidism on a stable dose of thyroid replacement therapy for at least three months prior to screening, and who have a screening thyroid-stimulating hormone within the limits of normal may participate)
* Has qualitative changes in lifestyle that, in the opinion of the investigator, would affect the subject's weight or disease status
* Had previous use of insulin within one month prior to screening, or more than seven total days of insulin treatment within three months prior to screening
* Has clinically significant cardiovascular and/or cerebrovascular disease including, but not limited to: 1) Previous history of stroke or transient ischemic attack, 2) Active, unstable coronary heart disease within the past six months, 3) Documented myocardial infarction within a year prior to screening 4) Any cardiac surgery including percutaneous transluminal coronary angioplasty or coronary artery bypass graft surgery within a year prior to screening 5) Unstable angina 6) Clinically significant arrhythmia or valvular heart disease within the past year 7) Congestive heart failure with New York Heart Association Class II to Class IV symptoms. Class I is acceptable. 8) Untreated hypertension, with systolic pressure greater than 160mm Hg and/or diastolic pressure greater than 95mm Hg. 9) ECG exclusion criteria: Heart rate is <40 and >110 beats per minute, PR Interval is <120 and >210msec, QRS duration is <70 and >120msec, QTc interval (Bazett) is >450msec or >480msec with bundle branch block
* Has fasting serum triglycerides ≥800mg/dL or 9mmol/L at screening (Visit 2). Subjects receiving lipid-lowering therapy must have been on the same dose of therapy for the past three months. Fasting is defined as no food/drink for at least eight hours prior to sampling
* If female, is currently lactating, pregnant, or actively trying to become pregnant
* Has significant renal disease as manifested by one or more of the following: 1) Creatinine clearance <60mL/min. (estimated from serum creatinine and demographic data using the modification of diet in renal disease calculation; refer to the SPM/ISFM), 2) Urine albumin excretion ≥500 µg/mL on a urine spot check, 3) Known loss of a kidney either by surgical ablation, injury, or disease
* Has history of significant comorbid diseases active within the last six months (e.g., gastrointestinal disease)
* Has history of pancreatitis within five years prior to randomization
* Has a documented history of chronic or advanced hepatobiliary disease including a history of, or positive laboratory results for, hepatitis at screening (Visit 2), and/or clinically significant hepatic enzyme elevation including: 1) Any two of the following enzymes greater than 1.5 times the upper limit of normal (ULN) value: - alanine aminotransferase (ALT), - aspartate aminotransferase (AST), - alkaline phosphatase (ALP), 2) Any one of the above enzymes two times greater than the ULN value AND total or direct bilirubin >1.5 times the ULN
* Has a history of alcohol or substance abuse within the past year, as determined by the investigator or a positive urine drug screen at screening (Visit 2) or during treatment: 1) Unwilling to refrain from the use of excessive alcohol or illicit drugs and adhere to other protocol-stated restrictions while participating in the study, 2) History of alcohol abuse defined as an average weekly intake of greater than 21 units or an average daily intake of greater than three units (males) or defined as an average weekly intake of greater than 14 units or an average daily intake of greater than two units (females). One unit is equivalent to a half-pint of beer or one measure of spirits or one glass of wine, 2) The investigator should exercise their medical judgment to determine if a urine drug screen is indicated
* Is currently taking prohibited concomitant medications listed in Section 6.6.2
* Has clinically significant anemia (i.e., hemoglobin <12.0g/dL or <120.0g/L for males and <11.0g/dL or <110.0g/L for females) or any other abnormal hematological profile that is considered by the investigator to be clinically significant
* Has known allergy to any formulation excipients, or history of drug or other allergy, which, in the opinion of the responsible study physician, contradicts participation
* Received treatment with an investigational drug or participated in any other clinical trial during the previous 30 days
* Has prior use of investigational agents with long half-lives of greater than seven days within the three months prior to screening
* Has any prior use of a GLP-1 analog, including GSK716155
* In the opinion of the investigator, has a risk of noncompliance with study procedures, or cannot read, understand, or complete study-related materials, particularly the informed consent
* Has any concurrent condition or any clinically significant abnormality identified on the screening physical examination, laboratory tests, ECG, including pulmonary, neurological, or inflammatory diseases, which, in the opinion of the investigator, may affect the interpretation of efficacy and safety data, or which otherwise, contraindicates participation in a clinical trial with a new chemical entity

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 361 (Actual)
Dates: Start 2007-04; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (149):
- United States (145):
  - GSK Investigational Site, Anniston, Alabama
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Bull Shoals, Arizona
  - GSK Investigational Site, Glendale, Arizona
  - GSK Investigational Site, Jonesboro, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Harrisburg, Arkansas
  - GSK Investigational Site, Jonesboro, Arkansas
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Searcy, Arkansas
  - GSK Investigational Site, Castro Valley, California
  - GSK Investigational Site, Culver City, California
  - GSK Investigational Site, Fullerton, California
  - GSK Investigational Site, Garden Grove, California
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Huntington Park, California
  - GSK Investigational Site, Lake Forest, California
  - GSK Investigational Site, Loma Linda, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Orange, California
  - GSK Investigational Site, Redwood City, California
  - GSK Investigational Site, Reedley, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, Van Buys, California
  - GSK Investigational Site, Ventura, California
  - GSK Investigational Site, Victorville, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Trumbull, Connecticut
  - GSK Investigational Site, Bradenton, Florida
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Gainesville, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Marianna, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Oviedo, Florida
  - GSK Investigational Site, Palm Harbor, Florida
  - GSK Investigational Site, Plantation, Florida
  - GSK Investigational Site, Tallahassee, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Winter Haven, Florida
  - GSK Investigational Site, Winter Park, Florida
  - GSK Investigational Site, Athens, Georgia
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Columbus, Georgia
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Perry, Georgia
  - GSK Investigational Site, Suwanee, Georgia
  - GSK Investigational Site, Tucker, Georgia
  - GSK Investigational Site, Honolulu, Hawaii
  - GSK Investigational Site, Meridian, Idaho
  - GSK Investigational Site, Aurora, Illinois
  - GSK Investigational Site, Evergreen Park, Illinois
  - GSK Investigational Site, La Grange, Illinois
  - GSK Investigational Site, Libertyville, Illinois
  - GSK Investigational Site, Oak Brook, Illinois
  - GSK Investigational Site, Watseka, Illinois
  - GSK Investigational Site, Anderson, Indiana
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, South Bend, Indiana
  - GSK Investigational Site, Ames, Iowa
  - GSK Investigational Site, Dubuque, Iowa
  - GSK Investigational Site, Kansas City, Kansas
  - GSK Investigational Site, Topeka, Kansas
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Covington, Louisiana
  - GSK Investigational Site, Lacombe, Louisiana
  - GSK Investigational Site, Metairie, Louisiana
  - GSK Investigational Site, Haverhill, Massachusetts
  - GSK Investigational Site, Caro, Michigan
  - GSK Investigational Site, Dearborn, Michigan
  - GSK Investigational Site, Kalamazoo, Michigan
  - GSK Investigational Site, Picayune, Mississippi
  - GSK Investigational Site, Rolling Fork, Mississippi
  - GSK Investigational Site, City of Saint Peters, Missouri
  - GSK Investigational Site, Jefferson City, Missouri
  - GSK Investigational Site, Springfield, Missouri
  - GSK Investigational Site, Billings, Montana
  - GSK Investigational Site, Lincoln, Nebraska
  - GSK Investigational Site, North Platte, Nebraska
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Buffalo, New York
  - GSK Investigational Site, Glens Falls, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Syracuse, New York
  - GSK Investigational Site, Williamsville, New York
  - GSK Investigational Site, Asheville, North Carolina
  - GSK Investigational Site, Chadbourn, North Carolina
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Mint Hill, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Wilmington, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Bismarck, North Dakota
  - GSK Investigational Site, Fargo, North Dakota
  - GSK Investigational Site, Grand Forks, North Dakota
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Toledo, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Bend, Oregon
  - GSK Investigational Site, Bensalem, Pennsylvania
  - GSK Investigational Site, Harrisburg, Pennsylvania
  - GSK Investigational Site, Morrisville, Pennsylvania
  - GSK Investigational Site, Uniontown, Pennsylvania
  - GSK Investigational Site, Watertown, South Dakota
  - GSK Investigational Site, Bristol, Tennessee
  - GSK Investigational Site, Clarksville, Tennessee
  - GSK Investigational Site, Johnson City, Tennessee
  - GSK Investigational Site, Knoxville, Tennessee
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, Milan, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Cleburne, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Euless, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, LaPorte, Texas
  - GSK Investigational Site, Lewisville, Texas
  - GSK Investigational Site, Longview, Texas
  - GSK Investigational Site, Midland, Texas
  - GSK Investigational Site, Missouri City, Texas
  - GSK Investigational Site, Pasadena, Texas
  - GSK Investigational Site, Pearland, Texas
  - GSK Investigational Site, Pharr, Texas
  - GSK Investigational Site, Round Rock, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, San Marcos, Texas
  - GSK Investigational Site, Spring, Texas
  - GSK Investigational Site, Sugar Land, Texas
  - GSK Investigational Site, The Woodlands, Texas
  - GSK Investigational Site, Tomball, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, South Burlington, Vermont
  - GSK Investigational Site, Chester, Virginia
  - GSK Investigational Site, Manassas, Virginia
  - GSK Investigational Site, Salem, Virginia
  - GSK Investigational Site, Madison, Washington
  - GSK Investigational Site, Spokane, Washington
- Chile (3):
  - GSK Investigational Site, Concepción, Región Del Biobio
  - GSK Investigational Site, Buin, Región Metro de Santiago
  - GSK Investigational Site, Santiago, Región Metro de Santiago
- GSK Investigational Site, Santo Domingo, Dominican Republic

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Rosenstock J, Reusch J, Bush M, Yang F, Stewart M; Albiglutide Study Group. Potential of albiglutide, a long-acting GLP-1 receptor agonist, in type 2 diabetes: a randomized controlled trial exploring weekly, biweekly, and monthly dosing. Diabetes Care. 2009 Oct;32(10):1880-6. doi: 10.2337/dc09-0366. Epub 2009 Jul 10. PMID 19592625
- [Derived] Young MA, Wald JA, Matthews JE, Scott R, Hodge RJ, Zhi H, Reinhardt RR. Clinical pharmacology of albiglutide, a GLP-1 receptor agonist. Postgrad Med. 2014 Nov;126(7):84-97. doi: 10.3810/pgm.2014.11.2836. PMID 25387217
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: GLP110125 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: GLP110125 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: GLP110125 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: GLP110125 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: GLP110125 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: GLP110125 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: GLP110125 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 361 participants were randomized into the study; however, only 356 of these participants received at least one dose of study drug.
Groups:
- Placebo: Participants received placebo weekly, administered as a subcutaneous injection for 16 weeks. Participants received subcutaneous injections alternating between the left and right sides of the body.
- Exenatide BID: Participants self-administered exenatide as a subcutaneous injection using prefilled pens, in accordance with current prescribing information. A dose of 5 micrograms (μg) was administered twice daily (BID) for the first 4 weeks, followed by a 12-week administration of a 10 μg BID dose. Participants who could not tolerate a 10 μg dose were to continue the study on the 5 μg BID dose.
- Albiglutide 4 mg Weekly: Participants received albiglutide 4 milligrams (mg) weekly, administered as a subcutaneous injection for 16 weeks. Participants received subcutaneous injections alternating between the left and right sides of the body.
- Albiglutide 15 mg Weekly: Participants received albiglutide 15 mg weekly, administered as a subcutaneous injection for 16 weeks. Participants received subcutaneous injections alternating between the left and right sides of the body.
- Albiglutide 30 mg Weekly: Participants received albiglutide 30 mg weekly, administered as a subcutaneous injection for 16 weeks. Participants received subcutaneous injections alternating between the left and right sides of the body.
- Albiglutide 15 mg Bi-weekly: Participants received albiglutide 15 mg every other week, alternating with placebo for each intervening week, administered as a subcutaneous injection for 16 weeks. Participants received subcutaneous injections alternating between the left and right sides of the body.
- Albiglutide 30 mg Bi-weekly: Participants received albiglutide 30 mg every other week, alternating with placebo for each intervening week, administered as a subcutaneous injection for 16 weeks. Participants received subcutaneous injections alternating between the left and right sides of the body.
- Albiglutide 50 mg Bi-weekly: Participants received albiglutide 50 mg every other week, alternating with placebo for each intervening week, administered as a subcutaneous injection for 16 weeks. Participants received subcutaneous injections alternating between the left and right sides of the body.
- Albiglutide 50 mg Every 4 Weeks: Participants received albiglutide 50 mg every 4 weeks, administered as a subcutaneous injection for 16 weeks. Participants received subcutaneous injections alternating between the left and right sides of the body.
- Albiglutide 100 mg Every 4 Weeks: Participants received albiglutide 100 mg every 4 weeks, administered as a subcutaneous injection for 16 weeks. Participants received subcutaneous injections alternating between the left and right sides of the body.
Period: Overall Study
Arm/Group | Placebo | Exenatide BID | Albiglutide 4 mg Weekly | Albiglutide 15 mg Weekly | Albiglutide 30 mg Weekly | Albiglutide 15 mg Bi-weekly | Albiglutide 30 mg Bi-weekly | Albiglutide 50 mg Bi-weekly | Albiglutide 50 mg Every 4 Weeks | Albiglutide 100 mg Every 4 Weeks
Started | 52 | 35 | 36 | 35 | 31 | 34 | 33 | 35 | 35 | 35
Safety Population | 51 (These participants received at least one dose of study drug.) | 35 (These participants received at least one dose of study drug.) | 35 (These participants received at least one dose of study drug.) | 35 (These participants received at least one dose of study drug.) | 31 (These participants received at least one dose of study drug.) | 33 (These participants received at least one dose of study drug.) | 32 (These participants received at least one dose of study drug.) | 35 (These participants received at least one dose of study drug.) | 35 (These participants received at least one dose of study drug.) | 34 (These participants received at least one dose of study drug.)
Completed | 40 | 29 | 19 | 24 | 21 | 19 | 25 | 20 | 30 | 20
Not Completed | 12 | 6 | 17 | 11 | 10 | 15 | 8 | 15 | 5 | 15
Not completed — Adverse Event | 6 | 1 | 5 | 6 | 5 | 5 | 5 | 10 | 2 | 9
Not completed — Lost to Follow-up | 0 | 0 | 2 | 3 | 1 | 3 | 0 | 1 | 1 | 1
Not completed — Protocol Violation | 1 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 5 | 0 | 2 | 1 | 0 | 2 | 1 | 3
Not completed — Lack of Efficacy | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Non-Compliance | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 1
Not completed — Treatment Eligibility Criteria Not Met | 1 | 1 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0
Not completed — Physician Prescribed Antidiabetic Drug | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Different Monotherapy Diabetic Drug | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Wrong Monotherapy Administered | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Violation of Exclusion Criteria | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Family Emergency; Had to Go to England | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrew Consent | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Moved Out of State | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Exenatide BID | Albiglutide 4 mg Weekly | Albiglutide 15 mg Weekly | Albiglutide 30 mg Weekly | Albiglutide 15 mg Bi-weekly | Albiglutide 30 mg Bi-weekly | Albiglutide 50 mg Bi-weekly | Albiglutide 50 mg Every 4 Weeks | Albiglutide 100 mg Every 4 Weeks | Total
Number analyzed (Participants) | 51 | 35 | 35 | 35 | 31 | 33 | 32 | 35 | 35 | 34 | 356
Age, Continuous [Mean (Standard Deviation); unit: Years] — Baseline data are reported for participants in the Safety Population, comprised of all randomly assigned participants who received at least one dose of study drug.
  Years | 54.0 (10.62) | 53.7 (9.38) | 50.4 (10.25) | 55.5 (10.48) | 54.2 (9.66) | 52.5 (9.55) | 55.5 (9.87) | 51.1 (10.25) | 54.1 (11.30) | 54.4 (9.89) | 53.5 (10.17)
Gender [Count of Participants; unit: Participants] — Baseline data are reported for participants in the Safety Population, comprised of all randomly assigned participants who received at least one dose of study drug.
  Participants
    Female | 23 | 19 | 20 | 17 | 23 | 19 | 16 | 16 | 18 | 15 | 186
    Male | 28 | 16 | 15 | 18 | 8 | 14 | 16 | 19 | 17 | 19 | 170
Race/Ethnicity, Customized [Number; unit: Participants] — Baseline data are reported for participants in the Safety Population, comprised of all randomly assigned participants who received at least one dose of study drug.
  Participants
    African American/African Heritage | 8 | 10 | 7 | 4 | 3 | 3 | 5 | 4 | 6 | 5 | 55
    American Indian or Alaskan Native | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 5
    Asian - Central/South Asian Heritage | 0 | 1 | 0 | 1 | 0 | 0 | 4 | 1 | 1 | 1 | 9
    Asian - East Asian Heritage | 2 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 8
    Asian - Japanese Heritage | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
    Asian - South East Asian Heritage | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 5
    Native Hawaiian or Other Pacific Islander | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 5
    White- Arabic/North African Heritage | 4 | 2 | 2 | 4 | 2 | 0 | 0 | 0 | 3 | 0 | 17
    White - White/Caucasian/European Heritage | 29 | 20 | 18 | 19 | 20 | 21 | 14 | 19 | 18 | 20 | 198
    Hispanic | 3 | 0 | 4 | 7 | 2 | 3 | 5 | 5 | 4 | 4 | 37
    Hispanic, Puerto Rican | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
    Mestizo | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 3
    Mexican | 3 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 8
    Mulatto | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 3
    Puerto Rican | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Week 16
Description: HbA1c is a form of hemoglobin that is measured primarily to identify the average plasma glucose concentration over a 2- to 3-month period. The Baseline HbA1c value is defined as the last non-missing value before the start of treatment. Change from Baseline in HbA1c was calculated as the value at Week 16 minus the value at Baseline. Based on ANCOVA: Change = treatment + Baseline HbA1c + prior therapy + gender + region. The last observation carried forward (LOCF) method was used to impute missing data, in which the last valid observation recorded on treatment (scheduled or unscheduled) was used to impute the missing measurement. For participants who had missing observations before their last observation on treatment, the closest previous non-missing on-treatment observation was carried forward to missing visits. If a participant had missing observation(s) immediately after Baseline, the Baseline observation was not carried forward and was left as missing.
Time Frame: Baseline and Week 16
Population: Intent-to-Treat (ITT) Population: all randomly assigned participants with at least one post-Baseline assessment of the primary endpoint. Participants from the exenatide arm were not included in the analysis. Only those participants with a value at Baseline and at the specified visit were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c in the blood
Arm/Group | Placebo | Exenatide BID | Albiglutide 4 mg Weekly | Albiglutide 15 mg Weekly | Albiglutide 30 mg Weekly | Albiglutide 15 mg Bi-weekly | Albiglutide 30 mg Bi-weekly | Albiglutide 50 mg Bi-weekly | Albiglutide 50 mg Every 4 Weeks | Albiglutide 100 mg Every 4 Weeks
Number analyzed (Participants) | 50 | 0 | 34 | 34 | 29 | 30 | 32 | 34 | 35 | 33
Percentage of HbA1c in the blood | -0.46 (0.136) |  | -0.25 (0.159) | -0.71 (0.160) | -1.08 (0.175) | -0.68 (0.167) | -1.01 (0.162) | -1.03 (0.159) | -0.80 (0.157) | -1.06 (0.161)
Statistical Analysis 1: Comparison: Placebo vs Albiglutide 4 mg Weekly; Test type: Superiority or Other; p = 0.2968, ANCOVA; Mean Difference (Final Values) = 0.20, 95% CI 2-sided [-0.18 to 0.59]
Statistical Analysis 2: Comparison: Placebo vs Albiglutide 15 mg Weekly; Test type: Superiority or Other; p = 0.1860, ANCOVA; Mean Difference (Final Values) = -0.26, 95% CI 2-sided [-0.64 to 0.12]
Statistical Analysis 3: Comparison: Placebo vs Albiglutide 30 mg Weekly; Test type: Superiority or Other; p = 0.0027, ANCOVA; Mean Difference (Final Values) = -0.62, 95% CI 2-sided [-1.03 to -0.22]
Statistical Analysis 4: Comparison: Placebo vs Albiglutide 15 mg Bi-weekly; Test type: Superiority or Other; p = 0.2766, ANCOVA; Mean Difference (Final Values) = -0.22, 95% CI 2-sided [-0.62 to 0.18]
Statistical Analysis 5: Comparison: Placebo vs Albiglutide 30 mg Bi-weekly; Test type: Superiority or Other; p = 0.0057, ANCOVA; Mean Difference (Final Values) = -0.55, 95% CI 2-sided [-0.94 to -0.16]
Statistical Analysis 6: Comparison: Placebo vs Albiglutide 50 mg Bi-weekly; Test type: Superiority or Other; p = 0.0032, ANCOVA; Mean Difference (Final Values) = -0.57, 95% CI 2-sided [-0.96 to -0.19]
Statistical Analysis 7: Comparison: Placebo vs Albiglutide 50 mg Every 4 Weeks; Test type: Superiority or Other; p = 0.0786, ANCOVA; Mean Difference (Final Values) = -0.34, 95% CI 2-sided [-0.72 to 0.04]
Statistical Analysis 8: Comparison: Placebo vs Albiglutide 100 mg Every 4 Weeks; Test type: Superiority or Other; p = 0.0022, ANCOVA; Mean Difference (Final Values) = -0.60, 95% CI 2-sided [-0.99 to -0.22]

2. Secondary Outcome: Change From Baseline in HbA1c at Weeks 4, 5, 7, 8, 9, 12, 15, and 16
Description: HbA1c is a form of hemoglobin that is measured primarily to identify the average plasma glucose concentration over a 2- to 3-month period. The Baseline HbA1c value is defined as the last non-missing value before the start of treatment. Change from Baseline in HbA1c was calculated as the post-Baseline value minus the value at Baseline. The last observation carried forward (LOCF) method was used to impute missing data, in which the last valid observation recorded on treatment (scheduled or unscheduled) was used to impute the missing measurement. For participants who had missing observations before their last observation on treatment, the closest previous non-missing on-treatment observation was carried forward to missing visits. If a participant had missing observation(s) immediately after Baseline, the Baseline observation was not carried forward and was left as missing.
Time Frame: Baseline and Weeks 4, 5, 7, 8, 9, 12, 15, and 16
Population: ITT Population. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles). Different participants may have been analyzed at different time points, so the overall number of participants analyzed reflects everyone in the ITT Population.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c in the blood
Arm/Group | Placebo | Exenatide BID | Albiglutide 4 mg Weekly | Albiglutide 15 mg Weekly | Albiglutide 30 mg Weekly | Albiglutide 15 mg Bi-weekly | Albiglutide 30 mg Bi-weekly | Albiglutide 50 mg Bi-weekly | Albiglutide 50 mg Every 4 Weeks | Albiglutide 100 mg Every 4 Weeks
Number analyzed (Participants) | 50 | 34 | 34 | 34 | 29 | 30 | 32 | 34 | 35 | 33
Percentage of HbA1c in the blood
  Week 4, n=47,34,33,34,28,29,31,34,34,30 | -0.14 (0.538) | -0.23 (0.485) | -0.12 (0.658) | -0.33 (0.442) | -0.56 (0.401) | -0.35 (0.470) | -0.34 (0.678) | -0.45 (0.547) | -0.41 (0.429) | -0.42 (0.523)
  Week 5, n=49,34,34,34,29,30,32,34,35,31 | -0.09 (0.570) | -0.32 (0.495) | -0.16 (0.758) | -0.39 (0.516) | -0.62 (0.439) | -0.42 (0.625) | -0.51 (0.756) | -0.58 (0.554) | -0.47 (0.608) | -0.65 (0.376)
  Week 7, n=50,34,34,34,29,30,32,34,35,32 | -0.15 (0.749) | -0.36 (0.554) | -0.19 (0.855) | -0.44 (0.619) | -0.79 (0.474) | -0.52 (0.648) | 0.64 (0.890) | -0.68 (0.831) | -0.45 (0.801) | -0.63 (0.420)
  Week 8, n=50,34,34,34,29,30,32,34,35,32 | -0.17 (0.793) | -0.45 (0.588) | -0.24 (0.897) | -0.50 (0.659) | -0.77 (0.494) | -0.54 (0.679) | -0.67 (0.928) | -0.71 (0.834) | -0.41 (0.823) | -0.68 (0.410)
  Week 9, n=50,34,34,34,29,30,32,34,35,32 | -0.21 (0.842) | -0.51 (0.633) | -0.19 (0.947) | -0.55 (0.713) | -0.85 (0.559) | -0.56 (0.767) | -0.71 (0.929) | -0.77 (0.842) | -0.54 (0.836) | -0.82 (0.486)
  Week 12, n=50,34,34,34,29,30,32,34,35,33 | -0.19 (0.892) | -0.56 (0.868) | -0.18 (1.025) | -0.58 (0.813) | -0.96 (0.649) | -0.59 (0.913) | -0.71 (1.003) | -0.79 (0.852) | -0.51 (0.942) | -0.84 (0.744)
  Week 15, n=50,34,34,34,29,30,32,34,35,33 | -0.27 (0.948) | -0.53 (0.865) | -0.19 (0.989) | -0.49 (0.819) | -0.86 (0.607) | -0.61 (0.929) | -0.79 (1.044) | -0.80 (1.041) | -0.58 (1.016) | -0.88 (0.790)
  Week 16, n=50,34,34,34,29,30,32,34,35,33 | -0.17 (1.006) | -0.54 (0.906) | -0.11 (1.156) | -0.49 (0.740) | -0.87 (0.652) | -0.56 (0.971) | -0.79 (0.978) | -0.79 (1.036) | -0.55 (1.012) | -0.87 (0.866)

3. Secondary Outcome: Number of Participants Who Achieved Target Values for HbA1c <6.5% and >=6.5% to <7% at Weeks 4, 5, 7, 8, 9, 12, 15, and 16
Description: The number of participants who achieved target values for HbA1c (i.e., HbA1c <6.5% and >=6.5% to <7%) were assessed. The last observation carried forward (LOCF) method was used to impute missing data, in which the last valid observation recorded on treatment (scheduled or unscheduled) was used to impute the missing measurement. For participants who had missing observations before their last observation on treatment, the closest previous non-missing on-treatment observation was carried forward to missing visits. If a participant had missing observation(s) immediately after Baseline, the Baseline observation was not carried forward and was left as missing.
Time Frame: Weeks (W) 4, 5, 7, 8, 9, 12, 15, and 16
Population: ITT Population. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles). Different participants may have been analyzed for different parameters at different time points, so the overall number of participants analyzed reflects everyone in the ITT Population.
Measure: Number; unit: Participants
Arm/Group | Placebo | Exenatide BID | Albiglutide 4 mg Weekly | Albiglutide 15 mg Weekly | Albiglutide 30 mg Weekly | Albiglutide 15 mg Bi-weekly | Albiglutide 30 mg Bi-weekly | Albiglutide 50 mg Bi-weekly | Albiglutide 50 mg Every 4 Weeks | Albiglutide 100 mg Every 4 Weeks
Number analyzed (Participants) | 50 | 34 | 34 | 34 | 29 | 30 | 32 | 34 | 35 | 33
Participants
  W4: <6.5%, n=47,34,33,34,28,29,31,34,34,30 | 1 | 0 | 0 | 1 | 4 | 0 | 0 | 3 | 1 | 3
  W4: >=6.5% to <7%, n=47,34,33,34,28,29,31,34,34,30 | 8 | 5 | 5 | 8 | 8 | 6 | 8 | 5 | 6 | 6
  W5: <6.5%, n=49,34,34,34,29,30,32,34,35,31 | 2 | 0 | 1 | 2 | 4 | 1 | 1 | 2 | 1 | 4
  W5: >=6.5% to <7%, n=49,34,34,34,29,30,32,34,35,31 | 4 | 7 | 5 | 7 | 8 | 5 | 9 | 11 | 7 | 12
  W7: <6.5%, n=50,34,34,34,29,30,32,34,35,32 | 1 | 1 | 1 | 4 | 8 | 1 | 3 | 6 | 2 | 5
  W7: >=6.5% to <7%, n=50,34,34,34,29,30,32,34,35,32 | 9 | 9 | 4 | 4 | 5 | 9 | 11 | 9 | 8 | 8
  W8: <6.5%, n=50,34,34,34,29,30,32,34,35,32 | 1 | 2 | 1 | 4 | 6 | 1 | 4 | 7 | 2 | 5
  W8: >=6.5% to <7%, n=50,34,34,34,29,30,32,34,35,32 | 10 | 7 | 6 | 8 | 8 | 9 | 12 | 10 | 4 | 11
  W9: <6.5%, n=50,34,34,34,29,30,32,34,35,32 | 3 | 2 | 2 | 6 | 8 | 1 | 3 | 7 | 2 | 9
  W9: >=6.5% to <7%, n=50,34,34,34,29,30,32,34,35,32 | 9 | 9 | 5 | 7 | 5 | 10 | 11 | 10 | 9 | 8
  W12: <6.5%, n=50,34,34,34,29,30,32,34,35,33 | 3 | 3 | 2 | 5 | 11 | 3 | 3 | 8 | 2 | 7
  W12:>=6.5% to <7%, n=50,34,34,34,29,30,32,34,35,33 | 7 | 8 | 4 | 8 | 5 | 7 | 13 | 11 | 9 | 8
  W15: <6.5%, n=50,34,34,34,29,30,32,34,35,33 | 3 | 4 | 2 | 4 | 8 | 4 | 6 | 10 | 3 | 9
  W15:>=6.5% to <7%, n=50,34,34,34,29,30,32,34,35,33 | 8 | 6 | 5 | 8 | 7 | 7 | 8 | 9 | 8 | 7
  W16: <6.5%, n=50,34,34,34,29,30,32,34,35,33 | 2 | 4 | 3 | 4 | 10 | 5 | 4 | 10 | 3 | 8
  W16:>=6.5% to <7%, n=50,34,34,34,29,30,32,34,35,33 | 8 | 8 | 3 | 8 | 5 | 3 | 12 | 8 | 5 | 8

4. Secondary Outcome: Change From Baseline in Waist Circumference at Week 16
Description: The Baseline value is the last non-missing value before the start of treatment. Change from Baseline in waist circumference was calculated as the value at Week 16 minus the value at Baseline. The last observation carried forward (LOCF) method was used to impute missing data, in which the last valid observation recorded on treatment (scheduled or unscheduled) was used to impute the missing measurement. For participants who had missing observations before their last observation on treatment, the closest previous non-missing on-treatment observation was carried forward to missing visits. If a participant had missing observation(s) immediately after Baseline, the Baseline observation was not carried forward and was left as missing.
Time Frame: Baseline and Week 16
Population: ITT Population. Only participants with a value at Baseline and at Week 16 were analyzed.
Measure: Mean (Standard Deviation); unit: Centimeters
Arm/Group | Placebo | Exenatide BID | Albiglutide 4 mg Weekly | Albiglutide 15 mg Weekly | Albiglutide 30 mg Weekly | Albiglutide 15 mg Bi-weekly | Albiglutide 30 mg Bi-weekly | Albiglutide 50 mg Bi-weekly | Albiglutide 50 mg Every 4 Weeks | Albiglutide 100 mg Every 4 Weeks
Number analyzed (Participants) | 50 | 34 | 34 | 34 | 29 | 30 | 32 | 34 | 35 | 33
Centimeters | -0.51 (3.847) | -3.53 (8.532) | -1.50 (3.902) | -3.16 (6.901) | -1.14 (3.856) | -1.83 (3.392) | -0.47 (3.589) | -2.00 (5.454) | -0.88 (5.146) | -0.77 (4.161)

5. Secondary Outcome: Change From Baseline in Body Weight at Week 16
Description: The Baseline value is the last non-missing value before the start of treatment. Change from Baseline in body weight was calculated as the value at Week 16 minus the value at Baseline. The last observation carried forward (LOCF) method was used to impute missing data, in which the last valid observation recorded on treatment (scheduled or unscheduled) was used to impute the missing measurement. For participants who had missing observations before their last observation on treatment, the closest previous non-missing on-treatment observation was carried forward to missing visits. If a participant had missing observation(s) immediately after Baseline, the Baseline observation was not carried forward and was left as missing.
Time Frame: Baseline and Week 16
Population: ITT Population. Only participants with a value at Baseline and at Week 16 were analyzed.
Measure: Mean (Standard Deviation); unit: Kilograms (Kg)
Arm/Group | Placebo | Exenatide BID | Albiglutide 4 mg Weekly | Albiglutide 15 mg Weekly | Albiglutide 30 mg Weekly | Albiglutide 15 mg Bi-weekly | Albiglutide 30 mg Bi-weekly | Albiglutide 50 mg Bi-weekly | Albiglutide 50 mg Every 4 Weeks | Albiglutide 100 mg Every 4 Weeks
Number analyzed (Participants) | 50 | 34 | 34 | 34 | 29 | 30 | 32 | 34 | 35 | 33
Kilograms (Kg) | -0.71 (2.883) | -2.41 (3.527) | -0.91 (1.733) | -0.90 (2.901) | -1.43 (2.371) | -1.76 (2.828) | -1.59 (2.455) | -1.14 (2.872) | -1.08 (3.177) | -1.65 (3.570)

6. Secondary Outcome: Percent Change From Baseline in Body Weight at Week 16
Description: The Baseline value is the last non-missing value before the start of treatment. Change from Baseline in body weight was calculated as the value at Week 16 minus the value at Baseline. Percent change from Baseline was calculated as the ([value at Week 16 minus the Baseline value] divided by the Baseline value) multiplied by 100. The LOCF method was used to impute missing data, in which the last valid observation recorded on treatment (scheduled or unscheduled) was used to impute the missing measurement. For participants who had missing observations before their last observation on treatment, the closest previous non-missing on-treatment observation was carried forward to missing visits. If a participant had missing observation(s) immediately after Baseline, the Baseline observation was not carried forward and was left as missing.
Time Frame: Baseline and Week 16
Population: ITT Population. Only participants with a value at Baseline and at Week 16 were analyzed.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo | Exenatide BID | Albiglutide 4 mg Weekly | Albiglutide 15 mg Weekly | Albiglutide 30 mg Weekly | Albiglutide 15 mg Bi-weekly | Albiglutide 30 mg Bi-weekly | Albiglutide 50 mg Bi-weekly | Albiglutide 50 mg Every 4 Weeks | Albiglutide 100 mg Every 4 Weeks
Number analyzed (Participants) | 50 | 34 | 34 | 34 | 29 | 30 | 32 | 34 | 35 | 33
Percent change | -0.72 (3.403) | -2.53 (4.307) | -0.94 (1.838) | -1.04 (3.261) | -1.59 (2.663) | -1.97 (2.908) | -1.69 (2.773) | -1.32 (3.160) | -1.37 (3.571) | -1.89 (3.190)

7. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Weeks 4, 5, 7, 8, 9, 12, 15, and 16
Description: The FPG test measures blood sugar levels after the participant has not eaten (fasted) for at least eight hours prior to the sampling. The Baseline FPG value is the last non-missing value before the start of treatment. Change from Baseline in FPG was calculated as the post-Baseline value minus the Baseline value. The LOCF method was used to impute missing data, in which the last valid observation recorded on treatment (scheduled or unscheduled) was used to impute the missing measurement. For participants who had missing observations before their last observation on treatment, the closest previous non-missing on-treatment observation was carried forward to missing visits. If a participant had missing observation(s) immediately after Baseline, the Baseline observation was not carried forward and was left as missing.
Time Frame: Baseline and Weeks 4, 5, 7, 8, 9, 12, 15, and 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Placebo | Exenatide BID | Albiglutide 4 mg Weekly | Albiglutide 15 mg Weekly | Albiglutide 30 mg Weekly | Albiglutide 15 mg Bi-weekly | Albiglutide 30 mg Bi-weekly | Albiglutide 50 mg Bi-weekly | Albiglutide 50 mg Every 4 Weeks | Albiglutide 100 mg Every 4 Weeks
Number analyzed (Participants) | 50 | 34 | 34 | 34 | 29 | 30 | 32 | 34 | 35 | 33
Millimoles per liter (mmol/L)
  Week 4, n=47,33,32,32,29,28,32,32,34,32 | -0.40 (2.565) | -1.11 (1.953) | -0.99 (3.037) | -0.58 (1.693) | -1.39 (1.968) | -1.06 (2.110) | -0.97 (1.629) | -1.35 (2.533) | -0.14 (3.192) | -0.61 (2.267)
  Week 5, n=47,33,32,32,29,28,32,32,34,32 | -0.40 (2.774) | -1.06 (2.377) | -1.02 (2.964) | -1.05 (1.705) | -1.53 (1.898) | -1.41 (2.363) | -1.72 (1.933) | -2.17 (2.453) | -1.55 (3.032) | -2.12 (1.959)
  Week 7, n=47,33,32,32,29,28,32,32,34,33 | -0.19 (2.924) | -1.25 (2.204) | -0.80 (2.942) | -0.13 (2.261) | -1.54 (1.723) | -1.16 (2.651) | -1.51 (2.065) | -1.87 (2.801) | -0.41 (2.844) | -1.07 (2.519)
  Week 8, n=47,33,32,32,29,28,32,32,34,33 | -0.44 (2.689) | -1.43 (2.258) | -1.22 (2.958) | -0.80 (1.856) | -1.60 (1.925) | -1.29 (2.520) | -1.27 (2.092) | -1.29 (2.655) | -0.66 (2.202) | -1.29 (2.898)
  Week 9, n=47,33,32,32,29,28,32,32,34,33 | -0.25 (3.185) | -1.54 (2.044) | -1.13 (2.915) | -0.71 (1.674) | -1.49 (2.122) | -1.29 (2.617) | -1.64 (2.505) | -1.68 (3.012) | -1.48 (2.887) | -2.25 (2.388)
  Week 12, n=47,33,32,32,29,28,32,32,34,33 | -0.27 (2.833) | -1.32 (2.518) | -1.04 (2.863) | -0.70 (2.413) | -1.85 (1.722) | -1.11 (2.492) | -1.57 (2.196) | -1.49 (2.908) | -0.49 (3.103) | -1.50 (3.310)
  Week 15, n=47,33,32,32,29,28,32,32,34,33 | -0.44 (2.733) | -1.27 (2.343) | -0.67 (2.984) | -0.70 (1.755) | -1.54 (1.680) | -1.45 (2.320) | -1.71 (2.133) | -1.66 (3.662) | -0.79 (2.757) | -1.27 (3.502)
  Week 16, n=47,33,32,32,29,28,32,32,34,33 | -0.10 (2.895) | -0.80 (2.482) | -0.47 (3.118) | -0.72 (1.683) | -1.44 (2.027) | -1.28 (2.427) | -1.58 (2.059) | -1.32 (3.523) | -0.72 (2.765) | -1.22 (3.497)

8. Secondary Outcome: Change From Baseline in Fasting Fructosamine at Weeks 5, 8, 12, and 16
Description: Fasting fructosamine levels were measured after the participant had not eaten (fasted) for at least eight hours prior to the sampling. The Baseline fructosamine value is the last non-missing value before the start of treatment. Change from Baseline in fructosamine was calculated as the post-Baseline value minus the Baseline value. The LOCF method was used to impute missing data, in which the last valid observation recorded on treatment (scheduled or unscheduled) was used to impute the missing measurement. For participants who had missing observations before their last observation on treatment, the closest previous non-missing on-treatment observation was carried forward to missing visits. If a participant had missing observation(s) immediately after Baseline, the Baseline observation was not carried forward and was left as missing.
Time Frame: Baseline and Weeks 5, 8, 12, and 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Micromoles per liter (µmol/L)
Arm/Group | Placebo | Exenatide BID | Albiglutide 4 mg Weekly | Albiglutide 15 mg Weekly | Albiglutide 30 mg Weekly | Albiglutide 15 mg Bi-weekly | Albiglutide 30 mg Bi-weekly | Albiglutide 50 mg Bi-weekly | Albiglutide 50 mg Every 4 Weeks | Albiglutide 100 mg Every 4 Weeks
Number analyzed (Participants) | 50 | 34 | 34 | 34 | 29 | 30 | 32 | 34 | 35 | 33
Micromoles per liter (µmol/L)
  Week 5, n=48,34,32,33,28,29,32,34,35,29 | -8.3 (38.68) | -24.7 (38.65) | -11.9 (50.55) | -23.8 (20.74) | -30.7 (31.28) | -21.3 (36.67) | -34.4 (41.71) | -30.1 (41.75) | -29.2 (46.57) | -32.5 (32.40)
  Week 8, n=50,34,33,34,28,29,32,34,35,31 | -10.1 (41.37) | -30.6 (32.47) | -13.1 (50.64) | -25.7 (31.34) | -35.5 (26.97) | -28.9 (42.46) | -40.9 (43.73) | -32.7 (42.44) | -24.9 (40.03) | -29.5 (49.98)
  Week 12, n=50,34,33,34,28,29,32,34,35,33 | -11.2 (41.61) | -30.1 (35.78) | -12.5 (55.41) | -26.7 (30.61) | -31.8 (35.07) | -25.2 (46.21) | -40.2 (43.37) | -32.7 (48.01) | -26.4 (46.85) | -31.1 (52.14)
  Week 16, n=50,34,33,34,28,29,32,34,35,33 | -3.2 (46.33) | -24.6 (41.88) | -7.8 (56.38) | -18.2 (28.01) | -30.8 (31.05) | -23.0 (49.58) | -38.1 (43.17) | -29.4 (56.23) | -26.5 (40.27) | -24.9 (49.08)

9. Secondary Outcome: Change From Baseline in Fasting C-peptide at Weeks 5, 8, 12, and 16
Description: Fasting C-peptide levels were measured after the participant had not eaten (fasted) for at least eight hours prior to the sampling. The Baseline C-peptide value is the last non-missing value before the start of treatment. Change from Baseline in C-peptide was calculated as the post-Baseline value minus the Baseline value. The LOCF method was used to impute missing data, in which the last valid observation recorded on treatment (scheduled or unscheduled) was used to impute the missing measurement. For participants who had missing observations before their last observation on treatment, the closest previous non-missing on-treatment observation was carried forward to missing visits. If a participant had missing observation(s) immediately after Baseline, the Baseline observation was not carried forward and was left as missing.
Time Frame: Baseline and Weeks 5, 8, 12, and 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Nanomoles per liter (nmol/L)
Arm/Group | Placebo | Exenatide BID | Albiglutide 4 mg Weekly | Albiglutide 15 mg Weekly | Albiglutide 30 mg Weekly | Albiglutide 15 mg Bi-weekly | Albiglutide 30 mg Bi-weekly | Albiglutide 50 mg Bi-weekly | Albiglutide 50 mg Every 4 Weeks | Albiglutide 100 mg Every 4 Weeks
Number analyzed (Participants) | 50 | 34 | 34 | 34 | 29 | 30 | 32 | 34 | 35 | 33
Nanomoles per liter (nmol/L)
  Week 5, n=48,33,32,33,27,28,32,33,35,30 | 0.004 (0.4464) | 0.274 (0.7431) | -0.020 (0.3374) | -0.034 (0.6149) | 0.089 (0.3459) | 0.015 (0.3782) | -0.128 (0.6990) | 0.004 (0.4130) | 0.072 (0.4130) | 0.230 (0.3595)
  Week 8, n=50,34,33,34,28,29,32,33,35,31 | -0.019 (0.4044) | 0.104 (0.4643) | -0.073 (0.2813) | -0.026 (0.6237) | 0.095 (0.5520) | -0.038 (0.3931) | -0.015 (0.7842) | -0.062 (0.3735) | 0.031 (0.4738) | 0.007 (0.3363)
  Week 12, n=50,34,33,34,28,29,32,33,35,33 | -0.092 (0.4264) | 0.174 (0.5445) | -0.044 (0.3426) | -0.046 (0.5904) | 0.023 (0.3698) | -0.098 (0.3773) | -0.153 (0.6463) | -0.076 (0.4458) | 0.155 (0.5257) | 0.062 (0.6038)
  Week 16, n=50,34,33,34,28,29,32,33,35,33 | -0.091 (0.3149) | 0.216 (0.6786) | -0.051 (0.3877) | -0.075 (0.6046) | 0.171 (0.4400) | -0.059 (0.4010) | -0.137 (0.6540) | -0.066 (0.4025) | 0.076 (0.5365) | -0.005 (0.4312)

10. Secondary Outcome: Change From Baseline in Fasting Glucagon at Weeks 5, 8, 12, and 16
Description: Fasting glucagon levels were measured after the participant had not eaten (fasted) for at least eight hours prior to the sampling. The Baseline glucagon value is the last non-missing value before the start of treatment. Change from Baseline in glucagon was calculated as the post-Baseline value minus the Baseline value. The LOCF method was used to impute missing data, in which the last valid observation recorded on treatment (scheduled or unscheduled) was used to impute the missing measurement. For participants who had missing observations before their last observation on treatment, the closest previous non-missing on-treatment observation was carried forward to missing visits. If a participant had missing observation(s) immediately after Baseline, the Baseline observation was not carried forward and was left as missing.
Time Frame: Baseline and Weeks 5, 8, 12, and 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Nanograms per liter (ng/L)
Arm/Group | Placebo | Exenatide BID | Albiglutide 4 mg Weekly | Albiglutide 15 mg Weekly | Albiglutide 30 mg Weekly | Albiglutide 15 mg Bi-weekly | Albiglutide 30 mg Bi-weekly | Albiglutide 50 mg Bi-weekly | Albiglutide 50 mg Every 4 Weeks | Albiglutide 100 mg Every 4 Weeks
Number analyzed (Participants) | 50 | 34 | 34 | 34 | 29 | 30 | 32 | 34 | 35 | 33
Nanograms per liter (ng/L)
  Week 5, n=48,33,33,33,27,28,32,34,35,30 | 3.8 (43.63) | -3.9 (39.26) | -3.2 (27.16) | -13.9 (29.05) | -3.6 (21.95) | -6.0 (26.83) | -7.6 (20.72) | -11.6 (29.48) | -9.3 (23.21) | 1.9 (30.27)
  Week 8, n=50,34,34,34,28,29,32,34,35,31 | 6.9 (49.05) | -14.8 (38.34) | -5.6 (22.91) | -15.6 (32.75) | -2.4 (17.78) | -12.4 (32.17) | -3.1 (22.64) | -10.7 (34.48) | -0.3 (41.71) | 0.5 (27.94)
  Week 12, n=50,34,34,34,28,29,32,34,35,33 | 0.1 (49.48) | -5.5 (32.41) | -8.6 (31.51) | -20.1 (36.53) | -4.5 (21.60) | -11.1 (39.08) | 0.2 (24.55) | -3.3 (35.85) | -3.7 (38.02) | -2.1 (23.58)
  Week 16, n=50,34,34,34,28,29,32,34,35,33 | -2.1 (45.73) | -4.5 (41.10) | -3.9 (26.72) | -20.5 (36.06) | -2.6 (22.70) | -7.1 (32.75) | -5.0 (17.95) | -10.9 (34.41) | -11.5 (25.21) | -4.7 (18.59)

11. Secondary Outcome: Change From Baseline in Fasting Insulin at Weeks 5, 8, 12, and 16
Description: Fasting insulin levels were measured after the participant had not eaten (fasted) for at least eight hours prior to the sampling. The Baseline insulin value is the last non-missing value before the start of treatment. Change from Baseline in insulin was calculated as the post-Baseline value minus the Baseline value. The LOCF method was used to impute missing data, in which the last valid observation recorded on treatment (scheduled or unscheduled) was used to impute the missing measurement. For participants who had missing observations before their last observation on treatment, the closest previous non-missing on-treatment observation was carried forward to missing visits. If a participant had missing observation(s) immediately after Baseline, the Baseline observation was not carried forward and was left as missing.
Time Frame: Baseline and Weeks 5, 8, 12, and 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Picomoles per liter (pmol/L)
Arm/Group | Placebo | Exenatide BID | Albiglutide 4 mg Weekly | Albiglutide 15 mg Weekly | Albiglutide 30 mg Weekly | Albiglutide 15 mg Bi-weekly | Albiglutide 30 mg Bi-weekly | Albiglutide 50 mg Bi-weekly | Albiglutide 50 mg Every 4 Weeks | Albiglutide 100 mg Every 4 Weeks
Number analyzed (Participants) | 50 | 34 | 34 | 34 | 29 | 30 | 32 | 34 | 35 | 33
Picomoles per liter (pmol/L)
  Week 5, n=47,31,32,33,27,28,31,30,33,30 | 5.1 (106.67) | 29.6 (104.29) | -12.4 (72.90) | -16.4 (114.61) | 0.4 (75.97) | 28.5 (99.26) | -38.3 (104.22) | -8.4 (75.38) | 11.1 (97.92) | 36.2 (115.31)
  Week 8, n=49,32,33,34,28,29,32,31,33,31 | 9.2 (106.05) | 5.4 (52.47) | -16.5 (64.88) | -8.5 (116.41) | 2.4 (98.07) | 18.6 (102.92) | -14.4 (104.76) | -16.8 (84.12) | 12.9 (92.97) | 6.6 (62.90)
  Week 12, n=49,32,33,34,28,29,32,31,33,33 | 8.8 (79.93) | 18.0 (60.31) | -12.4 (67.03) | -7.9 (106.19) | -1.1 (86.02) | 17.8 (99.18) | -26.1 (94.10) | 0.2 (90.27) | 38.0 (158.33) | 11.6 (73.33)
  Week 16, n=49,32,33,34,28,29,32,31,33,33 | -5.8 (42.74) | 17.4 (52.62) | 2.9 (81.64) | -19.9 (112.32) | 25.1 (114.95) | 21.9 (99.41) | -24.0 (90.05) | -17.4 (80.04) | 12.9 (72.22) | 18.4 (80.83)

12. Secondary Outcome: Change From Baseline in Triglycerides, Free Fatty Acids, Total Cholesterol, Low-density Lipoprotein Cholesterol, and High-density Lipoprotein Cholesterol at Weeks 5, 8, 12, and 16
Description: Serum lipid components, including triglycerides (TG), free fatty acids (FFA), total cholesterol (CL), low-density lipoprotein cholesterol (LDL-C), and high-density lipoprotein cholesterol (HDL-C), were measured at Baseline and Weeks 5, 8, 12, and 16. The Baseline value is the last non-missing value before the start of treatment. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. The LOCF method was used to impute missing data, in which the last valid observation recorded on treatment (scheduled or unscheduled) was used to impute the missing measurement. For participants who had missing observations before their last observation on treatment, the closest previous non-missing on-treatment observation was carried forward to missing visits. If a participant had missing observation(s) immediately after Baseline, the Baseline observation was not carried forward and was left as missing.
Time Frame: Baseline and Weeks 5, 8, 12, and 16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | Exenatide BID | Albiglutide 4 mg Weekly | Albiglutide 15 mg Weekly | Albiglutide 30 mg Weekly | Albiglutide 15 mg Bi-weekly | Albiglutide 30 mg Bi-weekly | Albiglutide 50 mg Bi-weekly | Albiglutide 50 mg Every 4 Weeks | Albiglutide 100 mg Every 4 Weeks
Number analyzed (Participants) | 50 | 34 | 34 | 34 | 29 | 30 | 32 | 34 | 35 | 33
mmol/L
  TG, Week 5, n=45,31,34,31,27,29,31,34,35,30 | -0.225 (1.0354) | -0.068 (0.7288) | 0.303 (2.1539) | -0.376 (1.1387) | 0.112 (0.6974) | -0.266 (1.2296) | -0.147 (1.0251) | -1.423 (3.7638) | -0.725 (1.3749) | -0.184 (0.5912)
  TG, Week 8, n=50,33,34,34,27,30,32,34,35,31 | -0.222 (1.5590) | -0.238 (0.6205) | 0.178 (2.1883) | -0.408 (1.3143) | -0.009 (0.6977) | -0.219 (1.0210) | -0.150 (0.9610) | -1.494 (3.8212) | -0.175 (1.6289) | -0.028 (1.1012)
  TG, Week 12, n=50,34,34,34,28,30,32,34,35,33 | -0.329 (1.2941) | 0.094 (1.4597) | 0.221 (2.3056) | -0.341 (1.2139) | 0.106 (0.8936) | -0.380 (0.8947) | -0.269 (1.0358) | -1.539 (3.9093) | -0.362 (1.5880) | 0.070 (0.8288)
  TG, Week 16, n=50,34,34,34,28,30,32,34,35,33 | -0.377 (1.6534) | -0.149 (0.8423) | 0.122 (2.1274) | -0.296 (1.2876) | 0.099 (0.9002) | -0.258 (0.9248) | -0.331 (0.9529) | -1.469 (3.8476) | -0.426 (1.7338) | -0.114 (1.1446)
  FFA, Week 5, n=48,33,32,33,27,28,32,34,35,29 | 0.029 (0.1867) | -0.038 (0.2518) | -0.032 (0.1691) | -0.008 (0.1392) | 0.014 (0.1381) | 0.025 (0.1927) | -0.028 (0.2017) | -0.012 (0.2266) | -0.001 (0.1568) | 0.006 (0.2237)
  FFA, Week 8, n=50,34,33,34,28,29,32,34,35,31 | 0.034 (0.2021) | -0.045 (0.2186) | 0.033 (0.1699) | -0.048 (0.1345) | 0.046 (0.1934) | 0.017 (0.1897) | -0.027 (0.1974) | -0.004 (0.2359) | 0.055 (0.1843) | 0.175 (0.8591)
  FFA, Week 12, n=50,34,33,34,28,29,32,34,35,33 | 0.075 (0.2018) | -0.007 (0.1882) | 0.022 (0.2003) | -0.013 (0.1870) | 0.043 (0.1826) | 0.010 (0.1920) | -0.051 (0.2250) | 0.011 (0.2481) | -0.030 (0.1796) | 0.123 (0.8347)
  FFA, Week 16, n=50,34,33,34,28,29,32,34,35,33 | 0.078 (0.2047) | -0.031 (0.1631) | 0.020 (0.2084) | 0.016 (0.2159) | 0.050 (0.1695) | 0.034 (0.2006) | -0.005 (0.2494) | 0.025 (0.2319) | 0.012 (0.2065) | 0.094 (0.8399)
  Total CL, Week 5, n=45,31,34,31,27,29,31,34,35,30 | -0.023 (0.6128) | -0.239 (0.6613) | -0.153 (0.8765) | -0.139 (0.5795) | -0.113 (0.6588) | -0.372 (0.6998) | -0.140 (0.4168) | -0.451 (0.9158) | -0.407 (0.6393) | -0.245 (0.5284)
  Total CL, Week 8, n=50,33,34,34,27,30,32,34,35,31 | -0.050 (0.5932) | -0.182 (0.6517) | -0.060 (0.9192) | -0.162 (0.4772) | 0.002 (0.5870) | -0.172 (0.6633) | -0.094 (0.4566) | -0.418 (0.8572) | -0.183 (0.8011) | 0.060 (0.6296)
  Total CL, Week 12, n=50,34,34,34,28,30,32,34,35,33 | 0.045 (0.6465) | 0.054 (0.7723) | -0.025 (0.9136) | -0.140 (0.5686) | -0.020 (0.6926) | -0.190 (0.5975) | -0.092 (0.8249) | -0.338 (0.9449) | -0.134 (0.6620) | 0.015 (0.5786)
  Total CL, Week 16, n=50,34,34,34,28,30,32,34,35,33 | 0.095 (0.7695) | -0.031 (0.8271) | -0.032 (0.9312) | -0.037 (0.5402) | 0.009 (0.5964) | -0.225 (0.5420) | -0.178 (0.4476) | -0.447 (0.8464) | -0.217 (0.7376) | 0.018 (0.5532)
  LDL-C, Week 5, n=41,29,31,29,26,28,29,27,32,29 | 0.066 (0.5417) | -0.153 (0.5479) | -0.294 (0.7053) | -0.155 (0.5653) | -0.068 (0.6225) | -0.285 (0.5345) | -0.082 (0.3708) | 0.026 (0.5064) | -0.106 (0.4576) | -0.091 (0.4910)
  LDL-C, Week 8, n=45,32,32,32,26,30,31,28,32,30 | 0.066 (0.5123) | -0.014 (0.5556) | -0.132 (0.7398) | -0.157 (0.5620) | 0.089 (0.6053) | -0.160 (0.5305) | -0.052 (0.4403) | 0.053 (0.4543) | -0.087 (0.4336) | 0.054 (0.5581)
  LDL-C, Week 12, n=45,33,32,32,28,30,31,28,32,32 | 0.138 (0.4923) | 0.105 (0.6259) | -0.096 (0.6483) | -0.152 (0.6477) | 0.004 (0.6456) | -0.034 (0.5547) | -0.004 (0.7153) | 0.156 (0.4614) | -0.061 (0.3790) | 0.010 (0.4771)
  LDL-C, Week 16, n=46,33,32,32,28,30,31,28,32,32 | 0.190 (0.6025) | 0.096 (0.6960) | -0.109 (0.6558) | -0.045 (0.6183) | 0.003 (0.6010) | -0.123 (0.5198) | -0.062 (0.3943) | 0.059 (0.5750) | -0.088 (0.5125) | 0.054 (0.4475)
  HDL-C, Week 5, n=45,31,34,31,27,29,31,34,35,30 | -0.020 (0.1189) | -0.047 (0.1420) | 0.001 (0.1203) | -0.010 (0.1491) | -0.063 (0.1425) | -0.038 (0.1215) | -0.045 (0.1434) | -0.076 (0.1553) | -0.047 (0.1765) | -0.053 (0.1129)
  HDL-C, Week 8, n=50,33,34,34,27,30,32,34,35,31 | -0.005 (0.1192) | -0.058 (0.1606) | 0.006 (0.1160) | 0.019 (0.1187) | -0.061 (0.1368) | -0.018 (0.1417) | -0.030 (0.1217) | -0.050 (0.1403) | -0.054 (0.1746) | -0.016 (0.1567)
  HDL-C, Week 12, n=50,34,34,34,28,30,32,34,35,33 | -0.011 (0.1341) | -0.003 (0.2269) | 0.004 (0.1258) | -0.019 (0.1115) | -0.061 (0.1674) | -0.018 (0.1323) | -0.041 (0.1998) | -0.029 (0.1303) | -0.033 (0.1445) | -0.045 (0.1411)
  HDL-C, Week 16, n=50,34,34,34,28,30,32,34,35,33 | -0.002 (0.1274) | -0.025 (0.2192) | -0.007 (0.1366) | -0.010 (0.1342) | -0.046 (0.1699) | -0.015 (0.1146) | -0.031 (0.1413) | -0.065 (0.1730) | -0.033 (0.1595) | -0.048 (0.1930)

13. Secondary Outcome: Change From Baseline in Functional Living Index - Emesis (FLIE) Scores at Week 16
Description: The FLIE questionnaire is used to record the participant's feelings/opinions concerning the effects of nausea/vomiting on their quality of life during the past five days. Participants completed the questionnaire by responding to 18 questions. The first set of 9 questions refer to nausea, and the second set of 9 questions refer to vomiting. Each question is scored on a seven-point visual analog scale (1 to 7). On this scale, a score of 1 corresponds to 0 millimeters (mm), and a score of 7 correspond to 100 mm. Anything in between is marked at the appropriate point on the scale and is measured in mm. Data are reported in mm in this table. In FLIE questions (FLIEQ) 1, 2, 4, 5, 7, 8, 9, 10, 12, 13, 14, 16, and 17, a score of 1 indicates no effect on the quality of life, and a score of 7 indicates a great effect on the quality of life. In FLIEQ 3, 6, 11, 15, and 18, a score of 1 indicates a great effect on the quality of life, and a score of 7 indicates no effect on the quality of life.
Time Frame: Baseline and Week 16
Population: Safety Population: all randomly assigned participants who received at least one dose of study drug. Only those participants available at the specified time point were analyzed. Change from Baseline was calculated as the score at Week 16 minus the score at Baseline.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Exenatide BID | Albiglutide 4 mg Weekly | Albiglutide 15 mg Weekly | Albiglutide 30 mg Weekly | Albiglutide 15 mg Bi-weekly | Albiglutide 30 mg Bi-weekly | Albiglutide 50 mg Bi-weekly | Albiglutide 50 mg Every 4 Weeks | Albiglutide 100 mg Every 4 Weeks
Number analyzed (Participants) | 37 | 28 | 19 | 25 | 22 | 19 | 24 | 21 | 29 | 22
Score on a scale
  FLIEQ1 | -0.1 (6.79) | -4.4 (19.25) | 5.7 (23.42) | 1.0 (19.54) | 4.6 (11.35) | 8.6 (24.35) | -1.0 (2.22) | 8.2 (22.66) | -0.3 (7.18) | -2.8 (8.30)
  FLIEQ2 | 0.2 (2.15) | -3.5 (18.64) | 5.5 (23.42) | 2.6 (18.20) | 3.0 (11.67) | 5.9 (22.87) | -0.8 (4.03) | 4.7 (21.95) | -0.6 (3.21) | -0.2 (1.84)
  FLIEQ3 | 15.6 (36.34) | 7.8 (25.52) | 10.3 (42.11) | -4.0 (19.64) | 18.6 (47.37) | 10.3 (45.34) | 3.9 (32.47) | 18.2 (39.83) | 4.5 (28.67) | 7.3 (29.72)
  FLIEQ4 | 0.4 (2.06) | -3.5 (18.32) | 6.4 (24.11) | -2.8 (11.95) | 1.5 (5.16) | 5.6 (22.91) | -1.6 (8.84) | 5.9 (22.48) | -1.9 (16.90) | -1.8 (6.68)
  FLIEQ5 | -0.3 (3.46) | -4.0 (18.21) | 6.4 (23.09) | -1.8 (7.18) | 2.9 (11.23) | 0.2 (33.34) | -1.3 (5.41) | 4.5 (21.97) | 1.5 (6.42) | -1.4 (6.03)
  FLIEQ6 | 11.2 (38.64) | 3.6 (29.76) | 9.4 (40.77) | -0.5 (26.11) | 20.0 (44.44) | 10.2 (45.38) | 4.2 (31.38) | 18.0 (40.06) | 5.6 (26.54) | 3.9 (36.69)
  FLIEQ7 | 0.4 (2.20) | -3.1 (19.16) | 5.7 (23.46) | 1.5 (16.77) | 0.2 (0.69) | 5.7 (22.88) | -1.0 (6.71) | 4.9 (21.93) | -0.1 (4.85) | -1.9 (6.44)
  FLIEQ8 | -0.6 (4.46) | -3.5 (18.60) | 5.7 (23.36) | -1.0 (10.95) | 2.6 (9.80) | 10.1 (29.33) | -0.7 (3.14) | 6.2 (22.05) | -0.4 (4.91) | -2.3 (7.08)
  FLIEQ9 | -0.1 (3.55) | -3.4 (17.86) | 5.3 (23.45) | -0.5 (3.64) | 2.3 (8.70) | 5.6 (22.91) | -0.7 (3.20) | 4.0 (22.33) | -0.1 (4.63) | -3.2 (9.80)
  FLIEQ10 | -0.3 (3.27) | -4.9 (18.81) | 5.8 (22.70) | -1.6 (6.51) | -0.1 (3.55) | 4.5 (23.37) | -0.3 (1.81) | 4.3 (22.00) | 0.2 (1.90) | -2.0 (5.12)
  FLIEQ11 | 15.3 (36.17) | 3.3 (30.36) | 13.8 (34.10) | -0.5 (38.39) | 21.9 (42.11) | 7.9 (46.96) | 3.6 (19.32) | 18.3 (40.27) | 7.2 (25.77) | 4.0 (36.47)
  FLIEQ12 | 0.1 (1.52) | -3.1 (17.45) | 6.4 (23.00) | -0.8 (8.09) | 1.8 (6.40) | 5.3 (22.95) | -0.2 (2.26) | 4.4 (21.97) | -0.4 (3.17) | -0.8 (3.49)
  FLIEQ13 | 0.1 (1.57) | -4.0 (18.31) | 6.3 (23.03) | -2.2 (8.43) | 1.0 (6.12) | 9.8 (29.41) | -0.3 (1.71) | 4.3 (22.02) | 0.0 (1.72) | -2.1 (6.55)
  FLIEQ14 | -0.3 (2.95) | -4.1 (18.18) | 6.4 (23.12) | -1.4 (6.22) | 1.8 (6.15) | 5.3 (22.94) | -0.1 (1.61) | 4.3 (22.0) | -0.1 (1.81) | -2.1 (6.36)
  FLIEQ15 | 15.5 (36.06) | 7.0 (23.57) | 14.2 (34.03) | -4.9 (18.87) | 19.7 (46.48) | 5.6 (50.36) | 3.5 (19.32) | 18.4 (40.22) | 1.5 (20.48) | 4.0 (36.71)
  FLIEQ16 | -0.4 (2.58) | -3.8 (18.20) | 6.3 (23.02) | -1.4 (7.37) | -0.5 (3.66) | 8.2 (25.92) | -0.1 (1.80) | 4.5 (21.95) | 0.9 (5.55) | -1.5 (4.32)
  FLIEQ17 | 0.1 (1.60) | -4.1 (18.14) | 6.3 (22.97) | -1.2 (6.08) | -1.2 (5.10) | 4.5 (23.36) | -0.2 (1.98) | 4.3 (22.02) | -1.1 (5.62) | -0.6 (3.89)
  FLIEQ18 | 18.1 (37.82) | 6.9 (23.47) | 14.2 (33.91) | -3.2 (17.62) | 14.9 (34.45) | 10.1 (45.39) | 7.1 (26.96) | 18.5 (40.09) | 5.7 (26.48) | 6.9 (30.76)

14. Secondary Outcome: Number of Participants With the Indicated Response to Questions on the Hunger, Craving, and Fullness Questionnaire (HCFQ) at Week 16
Description: The HCFQ questionnaire is used to record how often participants have felt hungry or craved food, and how full participants felt after finishing meals, on average, in the past week. Participants answered the following seven questions with the response that best described their feelings of hunger, craving, and fullness: Q1, "In the past week I was hungry"; Q2, "In the past week I thought about food"; Q3, "In the past week I wanted to eat"; Q4, "In the past week I ate more than I should have"; Q5, "In the past week, I craved specific food"; Q6, "In the past week when finished meals I felt full"; Q7, "In the past week when finished meals I felt satisfied."
Time Frame: Week 16
Population: Safety Population. Only those participants available at the specified time point were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | Exenatide BID | Albiglutide 4 mg Weekly | Albiglutide 15 mg Weekly | Albiglutide 30 mg Weekly | Albiglutide 15 mg Bi-weekly | Albiglutide 30 mg Bi-weekly | Albiglutide 50 mg Bi-weekly | Albiglutide 50 mg Every 4 Weeks | Albiglutide 100 mg Every 4 Weeks
Number analyzed (Participants) | 39 | 30 | 21 | 25 | 22 | 19 | 25 | 21 | 30 | 22
Participants
  Q1: Always | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 1
  Q1: Often | 5 | 5 | 2 | 7 | 6 | 3 | 5 | 2 | 6 | 6
  Q1: Sometimes | 28 | 17 | 15 | 14 | 14 | 8 | 17 | 11 | 20 | 12
  Q1: Rarely | 4 | 7 | 3 | 4 | 2 | 6 | 0 | 4 | 2 | 2
  Q1: Never | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 1
  Q2: Always | 1 | 1 | 0 | 0 | 0 | 1 | 3 | 2 | 3 | 2
  Q2: Often | 4 | 5 | 2 | 7 | 7 | 3 | 6 | 3 | 6 | 6
  Q2: Sometimes | 28 | 19 | 14 | 13 | 11 | 10 | 15 | 9 | 16 | 11
  Q2: Rarely | 5 | 4 | 5 | 5 | 4 | 4 | 0 | 4 | 4 | 2
  Q2: Never | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 3 | 1 | 1
  Q3: Always | 3 | 0 | 0 | 1 | 1 | 1 | 4 | 3 | 3 | 0
  Q3: Often | 7 | 5 | 4 | 4 | 7 | 4 | 4 | 2 | 6 | 9
  Q3: Sometimes | 26 | 20 | 16 | 18 | 13 | 10 | 16 | 12 | 17 | 11
  Q3: Rarely | 3 | 5 | 1 | 2 | 1 | 4 | 1 | 2 | 4 | 1
  Q3: Never | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
  Q4: Yes, definitely | 4 | 1 | 0 | 2 | 2 | 2 | 2 | 2 | 7 | 3
  Q4: Yes, probably | 15 | 8 | 8 | 9 | 9 | 9 | 12 | 5 | 9 | 12
  Q4: I don't know | 10 | 5 | 2 | 1 | 1 | 2 | 4 | 2 | 2 | 2
  Q4: Probably not | 7 | 12 | 10 | 9 | 7 | 4 | 4 | 5 | 10 | 4
  Q4: Definitely not | 3 | 4 | 1 | 4 | 3 | 2 | 3 | 7 | 2 | 1
  Q5: Always | 1 | 1 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0
  Q5: Often | 2 | 2 | 2 | 4 | 1 | 1 | 6 | 3 | 5 | 3
  Q5: Sometimes | 19 | 15 | 5 | 13 | 14 | 7 | 15 | 9 | 11 | 8
  Q5: Rarely | 16 | 8 | 11 | 4 | 5 | 8 | 2 | 6 | 9 | 8
  Q5: Never | 1 | 4 | 3 | 4 | 0 | 3 | 0 | 3 | 5 | 3
  Q6: Much too full | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 1
  Q6: Very full | 10 | 2 | 3 | 5 | 3 | 4 | 4 | 2 | 7 | 2
  Q6: Comfortably full | 26 | 28 | 18 | 17 | 18 | 13 | 20 | 18 | 18 | 17
  Q6: Slightly hungry | 3 | 0 | 0 | 2 | 1 | 2 | 0 | 0 | 2 | 2
  Q6: Very hungry | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Q7: Extremely satisfied | 3 | 0 | 1 | 1 | 1 | 0 | 2 | 1 | 2 | 1
  Q7: Satisfied | 27 | 27 | 17 | 17 | 19 | 15 | 22 | 15 | 23 | 14
  Q7: Neither satisfied nor dissatisfied | 9 | 3 | 3 | 5 | 1 | 3 | 1 | 5 | 4 | 5
  Q7: Dissatisfied | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 1 | 2
  Q7: Extremely dissatisfied | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

15. Secondary Outcome: Mean Clearance of Albiglutide
Description: Clearance is defined as the volume of plasma cleared of albiglutide per unit time. Samples were collected prior to the administration of study medication on dosing days (Weeks 0, 4, 5, 7, 8, 9, 12, 15) and on the day of the clinic visit at Weeks 16, 17, 18, 20, 23, and 27. The Week 5, 8, and 12 post-dose pharmacokinetic (PK) sampling was performed within 6 days of drug administration.
Time Frame: Weeks 0, 4, 5, 7, 8, 9, 12, 15, 16, 17 18, 20, 23, and 27
Population: PK Analysis Population: all participants for whom a PK sample was obtained and analyzed
Measure: Mean (95% Confidence Interval); unit: milliliters per hour
Groups:
- All Participants Receiving Any Dose of Albiglutide: Participants received one of the following doses of albiglutide: 4 mg weekly, 15 mg weekly, 30 mg weekly (administered as a subcutaneous injection for 16 weeks) ; 15 mg bi-weekly, 30 mg bi-weekly, 50 mg bi-weekly (alternating with placebo for each intervening week, administered as a subcutaneous injection for 16 weeks); 50 mg every 4 weeks, 100 mg every 4 weeks (administered as a subcutaneous injection for 16 weeks). Participants received subcutaneous injections alternating between the left and right sides of the body.
Arm/Group | All Participants Receiving Any Dose of Albiglutide
Number analyzed (Participants) | 267
milliliters per hour | 94.2 [90.1 to 98.9]

16. Secondary Outcome: Mean Volume of Distribution of Albiglutide
Description: Volume of distribution is defined as the apparent volume in which albiglutide is distributed. Samples were collected prior to the administration of study medication on dosing days (Weeks 0, 4, 5, 7, 8, 9, 12, 15) and on the day of the clinic visit at Weeks 16, 17, 18, 20, 23, and 27. The Week 5, 8, and 12 post-dose (PK sampling was performed within 6 days of drug administration.
Time Frame: Weeks 0, 4, 5, 7, 8, 9, 12, 15, 16, 17 18, 20, 23, and 27
Population: PK Analysis Population
Measure: Mean (95% Confidence Interval); unit: Liters
Arm/Group | All Participants Receiving Any Dose of Albiglutide
Number analyzed (Participants) | 267
Liters | 16400 [15600 to 17300]

17. Secondary Outcome: Mean Absorption Rate of Albiglutide
Description: Absorption rate is defined as the rate at which albiglutide enters the blood circulation. Samples were collected prior to the administration of study medication on dosing days (Weeks 0, 4, 5, 7, 8, 9, 12, 15) and on the day of the clinic visit at Weeks 16, 17, 18, 20, 23, and 27. The Week 5, 8, and 12 post-dose (PK sampling was performed within 6 days of drug administration.
Time Frame: Weeks 0, 4, 5, 7, 8, 9, 12, 15, 16, 17 18, 20, 23, and 27
Population: PK Analysis Population
Measure: Mean (95% Confidence Interval); unit: hour^-1
Arm/Group | All Participants Receiving Any Dose of Albiglutide
Number analyzed (Participants) | 267
hour^-1 | 0.0193 [0.017 to 0.022]

18. Secondary Outcome: Mean Half-maximal Effective Concentration (EC50) of Albiglutide for HbA1c and FPG
Description: EC50 is defined as the concentration of albiglutide that give a half-maximal HbA1c and FPG response. Samples were collected prior to the administration of study medication on dosing days (Weeks 0, 4, 5, 7, 8, 9, 12, 15) and on the day of the clinic visit at Weeks 16, 17, 18, 20, 23, and 27. The Week 5, 8, and 12 post-dose (PK sampling was performed within 6 days of drug administration. EC50 estimates used PK data as well as HbA1c and FPG efficacy data. EC50 was estimated from an inhibitory Emax (maximal possible effect of albiglutide) model.
Time Frame: Weeks 0, 4, 5, 7, 8, 9, 12, 15, 16, 17 18, 20, 23, and 27
Population: PK/PD Analysis Population: all participants in the PK Analysis Population with sufficient dosing history for inclusion in the PK/PD analysis
Measure: Mean (95% Confidence Interval); unit: nanograms per milliliter
Arm/Group | All Participants Receiving Any Dose of Albiglutide
Number analyzed (Participants) | 318
nanograms per milliliter
  HbA1c, Treatment-naïve group | 1140 [483 to 2990]
  HbA1c, Prior monotherapy group | 1230 [403 to 3560]
  FPG | 1970 [950 to 5410]

ADVERSE EVENTS:
Time Frame: On-therapy serious adverse events (SAEs) and non-serious AEs, defined as those that have a start date on or after the first day of study medication and within 56 days after the end of study medication, are reported.
Description: SAEs and non-serious AEs are reported for members of the Safety Population, comprised of all participants who received at least one dose of study treatment.
Arm/Group | Placebo | Exenatide BID | Albiglutide 4 mg Weekly | Albiglutide 15 mg Weekly | Albiglutide 30 mg Weekly | Albiglutide 15 mg Bi-weekly | Albiglutide 30 mg Bi-weekly | Albiglutide 50 mg Bi-weekly | Albiglutide 50 mg Every 4 Weeks | Albiglutide 100 mg Every 4 Weeks
Serious Adverse Events (participants affected / at risk) | 2/51 | 1/35 | 0/35 | 3/35 | 7/31 | 2/33 | 5/32 | 5/35 | 7/35 | 5/34
Other Adverse Events (participants affected / at risk) | 29/51 | 22/35 | 24/35 | 20/35 | 22/31 | 22/33 | 25/32 | 27/35 | 27/35 | 26/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=51) | Exenatide BID (N=35) | Albiglutide 4 mg Weekly (N=35) | Albiglutide 15 mg Weekly (N=35) | Albiglutide 30 mg Weekly (N=31) | Albiglutide 15 mg Bi-weekly (N=33) | Albiglutide 30 mg Bi-weekly (N=32) | Albiglutide 50 mg Bi-weekly (N=35) | Albiglutide 50 mg Every 4 Weeks (N=35) | Albiglutide 100 mg Every 4 Weeks (N=34)
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Prinzmetal angina (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Injection site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 1
Injection site hypersensitivity (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0
Injection site pruritus (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site rash (General disorders) | 0 | 0 | 0 | 2 | 2 | 0 | 1 | 2 | 0 | 0
Injection site reaction (General disorders) | 1 | 0 | 0 | 0 | 3 | 1 | 1 | 0 | 1 | 0
Injection site urticaria (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Nerve compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 (0) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=51) | Exenatide BID (N=35) | Albiglutide 4 mg Weekly (N=35) | Albiglutide 15 mg Weekly (N=35) | Albiglutide 30 mg Weekly (N=31) | Albiglutide 15 mg Bi-weekly (N=33) | Albiglutide 30 mg Bi-weekly (N=32) | Albiglutide 50 mg Bi-weekly (N=35) | Albiglutide 50 mg Every 4 Weeks (N=35) | Albiglutide 100 mg Every 4 Weeks (N=34)
Nausea (Gastrointestinal disorders) | 6 | 14 | 5 | 7 | 8 | 9 | 8 | 19 | 13 | 18
Vomiting (Gastrointestinal disorders) | 1 | 6 | 0 | 3 | 4 | 3 | 3 | 10 | 6 | 14
Diarrhoea (Gastrointestinal disorders) | 2 | 8 | 5 | 2 | 5 | 4 | 7 | 6 | 6 | 7
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 2 | 4
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 2 | 2 | 2 | 3 | 0 | 3
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0 | 1 | 1 | 4 | 1 | 2
Abdominal distension (Gastrointestinal disorders) | 2 | 0 | 1 | 1 | 1 | 0 | 3 | 2 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 2 | 1 | 2 | 1 | 0 | 2 | 2 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 1 | 4 | 0 | 1 | 0 | 1 | 0 | 0
Stomach discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 2 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 3 | 0 | 1 | 1 | 1 | 0 | 0 | 3
Nasopharyngitis (Infections and infestations) | 3 | 2 | 2 | 4 | 3 | 2 | 3 | 4 | 4 | 2
Urinary tract infection (Infections and infestations) | 3 | 0 | 2 | 2 | 1 | 0 | 0 | 1 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 5 | 4 | 3 | 0 | 3 | 5 | 2 | 1 | 3 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 3 | 3 | 2 | 3 | 3 | 0
Bronchitis (Infections and infestations) | 0 | 2 | 0 | 0 | 1 | 1 | 2 | 1 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 3 | 1 | 0 | 2 | 0
Headache (Nervous system disorders) | 3 | 4 | 6 | 5 | 5 | 6 | 5 | 4 | 5 | 8
Dizziness (Nervous system disorders) | 4 | 3 | 5 | 2 | 2 | 2 | 2 | 2 | 5 | 2
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 7 | 0 | 6 | 2 | 2 | 4 | 4 | 4 | 1 | 4
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 3 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 3 | 1 | 0 | 0 | 1 | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 5 | 2 | 2 | 2 | 2 | 2 | 2 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 4 | 2 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 3 | 0 | 1 | 0 | 2 | 1 | 0
Fatigue (General disorders) | 1 | 1 | 1 | 1 | 2 | 1 | 2 | 2 | 2 | 1
Injection site erythema (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 0 | 1
Injection site pruritus (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 2 | 0 | 1 | 3 | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 4 | 1 | 0 | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 2 | 1 | 0 | 1 | 1 | 1 | 1
Anxiety (Psychiatric disorders) | 1 | 1 | 1 | 1 | 0 | 1 | 3 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Hypertension (Vascular disorders) | 2 | 2 | 3 | 0 | 2 | 1 | 1 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Blood creatine phosphokinase increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Conjunctivitis (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.